CLINICAL TRIAL: NCT00471042
Title: Buprenorphine for Treatment of Opioid Dependence in Primary Care
Brief Title: Study of Buprenorphine Maintenance Treatment for Opioid Dependence in Primary Care
Status: Completed | Type: Observational
Sponsor: New York State Psychiatric Institute (Other)
Collaborators: National Institute on Drug Abuse (NIDA) (NIH)
Responsible Party: Principal Investigator, Frances R Levin, Director of Substance Use Disorder, New York State Psychiatric Institute
Other Study IDs: #5258; NIDA-020000; K23DA020000 (NIH)
Record Dates: First submitted 2007-05-07; First posted 2007-05-09 (Estimated); Last update posted 2019-04-23 (Actual); Status verified 2019-04

CONDITIONS: Heroin Dependence; Opioid-Related Disorders; Substance Abuse, Intravenous
Keywords: Heroin Dependence; Opioid Dependence; Primary Care; Buprenorphine
MeSH Terms: conditions — Heroin Dependence; Opioid-Related Disorders; Substance Abuse, Intravenous | interventions — Buprenorphine

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Drug: Buprenorphine — Dose is determined according to the participants' individual need.

SUMMARY:
The purpose of this treatment research study is to assess the effectiveness of buprenorphine maintenance treatment for opioid dependence delivered in a primary care clinic setting. This study will determine whether buprenorphine treatment in primary care is effective in reducing cravings, reducing illicit opioid use, reducing addiction severity, and retaining patients in primary care treatment for opioid dependence.

DETAILED DESCRIPTION:
Buprenorphine maintenance treatment of opioid dependence in primary care may expand treatment access. Buprenorphine is a partial mu-opioid agonist approved for treatment of opioid dependence (dependence on heroin, prescription opioid pain medication, or methadone), which can be prescribed in primary care by authorized physicians. The purpose of this study is to assess the effectiveness of buprenorphine maintenance treatment in a primary care setting. Outcome measures include illicit opioid use during treatment, addiction severity scores from the Addiction Severity Index (ASI), patient craving ratings on a 100mm visual analog scale (VAS), and patient retention in treatment.

This is a 6-month, prospective cohort study of adults aged 18-65 who are seeking buprenorphine maintenance treatment for opioid dependence. This study is observational, not experimental, and patients will be treated in a naturalistic condition according to their individual treatment needs. Clinic visits will occur weekly for the first 4 weeks (Induction and Stabilization Phases), and monthly for the remaining 20 weeks (Maintenance Phase), at which time up to a month of medication may be prescribed. Participation in ancillary psychosocial treatment is recommended but not required. Urine toxicology and craving ratings will be collected at each visit. Additionally, research visits will occur monthly to collect data assessing addiction severity, risk factors, general health, and psychiatric symptoms.

ELIGIBILITY:
Inclusion Criteria:

* DSM-IV criteria for current opioid dependence
* Must be seeking treatment
* Must describe opioid medication or heroin as primary drug of abuse
* Must be financially able to receive treatment at the primary care clinic site and to receive medication (e.g., Medicaid)
* Able to give informed consent and comply with study procedures

Exclusion Criteria:

* Axis I psychiatric disorder(s) as defined by DSM-IV-TR that are unstable or would be disrupted by study participation
* Individuals at significant risk for suicide based on current mental state
* DSM-IV dependence with physiologic dependence other than opioid and nicotine
* Women must not be pregnant or lactating, and must agree to use a proven effective method of contraception and not become pregnant during the study
* Unstable physical disorder that might make participation hazardous
* Known allergy, sensitivity or adverse reaction to buprenorphine
* Current buprenorphine maintenance
* Inability to read or understand the self-report assessment forms unaided

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adults aged 18-65 who are seeking buprenorphine maintenance treatment for opioid dependence
Sampling Method: Non-Probability Sample
Enrollment: 30 (Actual)
Dates: Start 2006-06; Primary Completion 2008-08 (Actual); Study Completion 2012-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Erik W. Gunderson, M.D., Principal Investigator — Columbia University
Locations (1):
- Columbia University/New York State Psychiatric Institute, New York, New York, United States